CLINICAL TRIAL: NCT02584738
Title: Efficacy of Nebulized Magnesium Sulfate as an Adjunct to Standard Therapy in Asthma Exacerbation. A Randomized Controlled Trial
Brief Title: Nebulized Magnesium Sulfate as an Adjunct to Standard Therapy in Asthma Exacerbation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HGNAE-03
Record Dates: First submitted 2015-10-14; First posted 2015-10-23 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: Asthma; Exacerbation; Nebulization; Magnesium; Pediatric
MeSH Terms: conditions — Asthma | interventions — Ipratropium; Methylprednisolone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulized Magnesium Sulfate (Experimental): Nebulized salbutamol and ipratropium bromide mixed with 2.5 ml of isotonic MgSO4.
  Intravenous methylprednisolone or oral prednisolone
  Interventions: Drug: Nebulized Magnesium Sulfate; Drug: Nebulized Salbutamol; Drug: Ipratropium bromide; Drug: Methylprednisolone or Prednisolone
- Nebulized isotonic saline (Placebo Comparator): Nebulized salbutamol and ipratropium bromide with 2.5 ml of isotonic saline. Intravenous methylprednisolone or oral prednisolone
  Interventions: Drug: Nebulized isotonic saline; Drug: Nebulized Salbutamol; Drug: Ipratropium bromide; Drug: Methylprednisolone or Prednisolone

INTERVENTIONS:
Drug: Nebulized Magnesium Sulfate — Nebulized salbutamol and ipratropium bromide mixed with 2.5 ml of isotonic MgSO4 (150 mg) per dose every 20 minutes during the first hour.
  will be continued with nebulized standard treatment every hour for 4 hours.
  Other Names: MgSO4
  Arms: Nebulized Magnesium Sulfate
Drug: Nebulized isotonic saline — Nebulized salbutamol and ipratropium bromide mixed with 2.5 ml of isotonic saline per dose every 20 minutes during the first hour.
  will be continued with nebulized standard treatment every hour for 4 hours.
  Other Names: Standard treatment
  Arms: Nebulized isotonic saline
Drug: Nebulized Salbutamol — Nebulized salbutamol 2.5mg (2-5 years) or 5 mg (≥6 years)
Drug: Ipratropium bromide — Nebulized ipratropium bromide 250 mcg
Drug: Methylprednisolone or Prednisolone — Begin with intravenous methylprednisolone or oral prednisolone 2 mg/kg/day for each treatment
  Other Names: Corticosteroid therapy

SUMMARY:
The purpose of this study is to investigate the effectiveness of nebulized magnesium sulfate in patient with moderate to severe asthma exacerbation in pediatric emergency

DETAILED DESCRIPTION:
The inclusion period of the patients in this research will be on September 2015 to November 2015. Patients are going to be selected by the medical staff on duty in the emergency paediatric service, according to the criteria previously established inclusion and exclusion. Immediately a baseline degree of respiratory distress using PRAM scale and heart rate, respiratory rate, blood pressure and oxygen saturation. While informed consent in which the objective and characteristics of the study will be obtained will be explained.

Patients will be randomly assigned one of the two treatments in the Research: standard treatment for moderate to severe asthma attack, according to GINA or standard treatment plus nebulised magnesium sulphate, according to the table of random allocation of treatment.

Evaluations were performed after administration of each spray, that is, at 20, 40, 60, 120, 180 and 240 minutes after beginning treatment. The parameters' to evaluate are going to be heart rate, respiratory rate, oxygen saturation, blood pressure and assessment of severity of acute asthma with PRAM scale.

The application of nebulized drugs are made in the emergency department of pediatrics by inhalation therapy staff who are also responsible for the preparation of medicines. It is clear that this staff not participate in the evaluation of patients, which will be performed by the research staff or by medical staff on duty in the pediatric emergency department.

Patients and evaluating physician will not pick out between the two solutions for nebulization not only colour but also smell or other special feature, because the solutions were arranged in two identical syringes. Administered alone at the end of the study treatment is known.

Later the entry or exit of the patient decide, who can be egress to show clinical improvement with decreased severity index PRAM, patients will be graduates of an outpatient treatment according to international guidelines on the management of acute asthma. All initial and outcome data will be recorded in a format of data collection All decisions will be made by patients pediatricians emergency department which will follow patients throughout the study and will have the power to release the study patients to use other interventions that they consider clinically necessary

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate or severe asthma exacerbations
* 2 to 15 years old.
* Served in the pediatric emergency department of naval high specialty General Hospital from September to December 2015.
* Signing the consent by the parents.

Exclusion Criteria:

* Coexistence of lung disease.
* Severe kidney disease.
* Severe liver disease.
* Pregnancy.
* Known previous reaction to magnesium.
* Parents who have not signed the agreement.
* Patients without a clinical history of asthma.
* Clinical diagnosis of mild asthma attack.
* Previously included in the study.
* Presence of comorbidities that endanger the patient's life.
* The patient has clinical or gasometric criteria for advanced airway management.
* Life-threatening symptoms.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 152 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Preschool Respiratory Assessment Measure (PRAM) | 20, 40, 60, 120, 180 and 240 minutes after beginning treatment
  Scalene muscle contraction, Suprasternal retractions, Wheezing, Air entry and O2 saturation.
  The score will be considering from the addition per each primary measure.
Change from Baseline Scalene muscle contraction | 20, 40, 60, 120, 180 and 240 minutes after beginning treatment
  Absent (0) or Present (2)
Change from Baseline Suprasternal retractions | 20, 40, 60, 120, 180 and 240 minutes after beginning treatment
  Absent (0) or Present (2)
Change from Baseline Wheezing | 20, 40, 60, 120, 180 and 240 minutes after beginning treatment
  Normal (0), Decreased at bases (1), Widespread decrease (2), or Absent/minimal (3)
Change from Baseline Air entry | 20, 40, 60, 120, 180 and 240 minutes after beginning treatment
  Absent (0), Expiratory only (1), Inspiratory and expiratory (2) or Audible without (3) stethoscope/silent chest with minimal air entry
Change from Baseline O2 saturation | 20, 40, 60, 120, 180 and 240 minutes after beginning treatment
  ≥95% (0), 92%-94% (1) or <92% (2)

SECONDARY OUTCOMES:
Rate of hospitalization | 4 hour
  Reduction the rate of hospitalization
Change from Baseline Heart rate | 20, 40, 60, 120, 180 and 240 minutes after beginning treatment
  Beats per minute
Change from Baseline Respiratory rate | 20, 40, 60, 120, 180 and 240 minutes after beginning treatment
  Breaths per minute
Change from Baseline Blood pressure | 60 minutes after beginning treatment
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Abisai Uicab Saucedo, Pediatrician, Principal Investigator — Secretaria de Marina
Locations (1):
- Hospital General Naval de Alta Especialidad, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Birken CS, Parkin PC, Macarthur C. Asthma severity scores for preschoolers displayed weaknesses in reliability, validity, and responsiveness. J Clin Epidemiol. 2004 Nov;57(11):1177-81. doi: 10.1016/j.jclinepi.2004.02.016. PMID 15567635
- [Background] Gorelick MH, Stevens MW, Schultz TR, Scribano PV. Performance of a novel clinical score, the Pediatric Asthma Severity Score (PASS), in the evaluation of acute asthma. Acad Emerg Med. 2004 Jan;11(1):10-8. doi: 10.1197/j.aem.2003.07.015. PMID 14709423
- [Background] Rodrigo GJ, Plaza Moral V, Forns SB, Castro-Rodriguez JA, de Diego Damia A, Cortes SL, Moreno CM, Nannini LJ, Neffen H, Salas J; SEPAR; ALAT. [ALERTA 2 guidelines. Latin America and Spain: recommendations for the prevention and treatment of asmatic exacerbations. Spanish Pulmonology and Thoracic Surgery Society (SEPAR). Asthma Department of the Latinamerican Thoracic Association (ALAT)]. Arch Bronconeumol. 2010 Oct;46 Suppl 7:2-20. doi: 10.1016/S0300-2896(10)70041-7. No abstract available. Spanish. PMID 21320808
- [Background] Gourgoulianis KI, Chatziparasidis G, Chatziefthimiou A, Molyvdas PA. Magnesium as a relaxing factor of airway smooth muscles. J Aerosol Med. 2001 Fall;14(3):301-7. doi: 10.1089/089426801316970259. PMID 11693841
- [Background] Dominguez LJ, Barbagallo M, Di Lorenzo G, Drago A, Scola S, Morici G, Caruso C. Bronchial reactivity and intracellular magnesium: a possible mechanism for the bronchodilating effects of magnesium in asthma. Clin Sci (Lond). 1998 Aug;95(2):137-42. PMID 9680494
- [Background] Cairns CB, Kraft M. Magnesium attenuates the neutrophil respiratory burst in adult asthmatic patients. Acad Emerg Med. 1996 Dec;3(12):1093-7. doi: 10.1111/j.1553-2712.1996.tb03366.x. PMID 8959161
- [Background] Mohammed S, Goodacre S. Intravenous and nebulised magnesium sulphate for acute asthma: systematic review and meta-analysis. Emerg Med J. 2007 Dec;24(12):823-30. doi: 10.1136/emj.2007.052050. PMID 18029512
- [Background] Shan Z, Rong Y, Yang W, Wang D, Yao P, Xie J, Liu L. Intravenous and nebulized magnesium sulfate for treating acute asthma in adults and children: a systematic review and meta-analysis. Respir Med. 2013 Mar;107(3):321-30. doi: 10.1016/j.rmed.2012.12.001. Epub 2013 Jan 3. PMID 23290189
- [Background] Powell C, Dwan K, Milan SJ, Beasley R, Hughes R, Knopp-Sihota JA, Rowe BH. Inhaled magnesium sulfate in the treatment of acute asthma. Cochrane Database Syst Rev. 2012 Dec 12;12:CD003898. doi: 10.1002/14651858.CD003898.pub5. PMID 23235599
- [Background] Goodacre S, Cohen J, Bradburn M, Gray A, Benger J, Coats T; 3Mg Research Team. Intravenous or nebulised magnesium sulphate versus standard therapy for severe acute asthma (3Mg trial): a double-blind, randomised controlled trial. Lancet Respir Med. 2013 Jun;1(4):293-300. doi: 10.1016/S2213-2600(13)70070-5. Epub 2013 May 17. PMID 24429154
- [Background] Powell CV, Kolamunnage-Dona R, Lowe J, Boland A, Petrou S, Doull I, Hood K, Williamson PR; MAGNETIC study group. MAGNEsium Trial In Children (MAGNETIC): a randomised, placebo-controlled trial and economic evaluation of nebulised magnesium sulphate in acute severe asthma in children. Health Technol Assess. 2013 Oct;17(45):v-vi, 1-216. doi: 10.3310/hta17450. PMID 24144222
- [Background] Alansari K, Ahmed W, Davidson BL, Alamri M, Zakaria I, Alrifaai M. Nebulized magnesium for moderate and severe pediatric asthma: A randomized trial. Pediatr Pulmonol. 2015 Dec;50(12):1191-9. doi: 10.1002/ppul.23158. Epub 2015 Feb 4. PMID 25652104
- [Background] Rowe BH. Intravenous and inhaled MgSO4 for acute asthma. Lancet Respir Med. 2013 Jun;1(4):276-7. doi: 10.1016/S2213-2600(13)70097-3. Epub 2013 May 17. No abstract available. PMID 24429139
- [Background] Petrou S, Boland A, Khan K, Powell C, Kolamunnage-Dona R, Lowe J, Doull I, Hood K, Williamson P. Economic evaluation of nebulized magnesium sulphate in acute severe asthma in children. Int J Technol Assess Health Care. 2014 Oct;30(4):354-60. doi: 10.1017/S0266462314000440. Epub 2014 Nov 14. PMID 25394502
- [Background] Wang H, Xiong Y, Gong C, Yin L, Yan L, Yuan X, Liu S, Shi T, Dai J. Effect of inhaled magnesium sulfate on bronchial hyperresponsiveness. Indian J Pediatr. 2015 Apr;82(4):321-7. doi: 10.1007/s12098-014-1476-6. Epub 2014 Jun 12. PMID 24916134
- [Result] Smith SR, Baty JD, Hodge D 3rd. Validation of the pulmonary score: an asthma severity score for children. Acad Emerg Med. 2002 Feb;9(2):99-104. doi: 10.1111/j.1553-2712.2002.tb00223.x. PMID 11825832
- [Result] Chalut DS, Ducharme FM, Davis GM. The Preschool Respiratory Assessment Measure (PRAM): a responsive index of acute asthma severity. J Pediatr. 2000 Dec;137(6):762-8. doi: 10.1067/mpd.2000.110121. PMID 11113831
- See also: Global Initiative for Asthma (GINA). Global strategy for asthma management and prevention (Updated 2015). — http://www.ginasthma.org